CLINICAL TRIAL: NCT01650766
Title: Study of S1 Efficacy and Toxicity as Second-line Treatment on Inoperable or Advanced Gastric Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Xu jianming, Director of Department of Digestive Oncology, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Other Study IDs: AGC-307PLAH-XJM
Record Dates: First submitted 2012-01-19; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The paraffin-embedded pathelogical tissues of tumors and the blood samples before and after medication are retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of the study is to investigate the correlation between the efficacy and toxicity of S-1 on gastric cancers and the expression of thymidylate synthase (TS), dihydropyrimidine dehydrogenase (DPD) and orotate phosphoribosyltransferase(OPRT).

DETAILED DESCRIPTION:
TS, DPD and OPRT are the key enzymes on the metabolic pathway of 5-Fu. We will retrospectively analyze the clinicopathological features of the patients who have suffered an inoperative or recurrent gastric cancers and administrated with S-1, such as the overall survival (OS), progressive-free survival (PFS), Lauren's classification and toxicity of S1, etc. We will divide the patients into several subgroups according to the parameters above, and then investigate the correlation between the parameters and the expression of TS, DPD and OPRT.

All of the analysis is retrospective, there is no different treatment operation once the subject enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, inoperable or advanced gastric cancer patients who received at most 1st line treatment
2. Aged 18 years or older
3. KPS performance status of ≥ 70.
4. Anticipated life expectancy of ≥ 3 months.
5. Adequate organ function, including bone marrow, kidney and liver.

   * ANC ≥ 1.5×109/L and hemoglobin ≥ 8g/dL and platelet count ≥ 100×109/L
   * Serum total bilirubin ≤ 1.5 x ULN, Serum ALT and AST ≤ 2.5 x ULN (Serum ALT and AST ≤ 5 x ULN, if liver metastases are present)
   * Serum creatinine ≤ 1.5 x ULN and CLcr > 60 ml/min
6. Written informed consent can be obtained prior to their participation in the trial.

Exclusion Criteria:

1. History of severe drug allergy , or an allergy to any components of S1
2. Subjects who have received chemotherapy, immunotherapy or radiotherapy within two weeks
3. Alimentary tract hemorrhage, diarrhea or aphagosis at the present stage
4. Subjects with uncontrolled CNS metastasis or epilepsia or severe psychiatric disorders.
5. Subjects who are regarded to be unsuitable for this trial by the investigator.
6. Subjects who are participating in other clinical trials
7. Subjects with ascites draining or severe infection
8. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with inoperable or advanced gastric cancers
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Jianming, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China